CLINICAL TRIAL: NCT02678767
Title: Ferumoxytol-enhanced Imaging and Quantitative Susceptibility Mapping in neuroAIDS
Brief Title: Ferumoxytol-enhanced Imaging and Mapping in neuroAIDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beau Nakamoto (Other)
Collaborators: Hawaii Pacific Health (Other); University of Hawaii (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Beau Nakamoto, Assistant Professor of Medicine, University of Hawaii
Organization: University of Hawaii (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2013-077; H032 (Other: Hawaii Center for AIDS); 1R21NS087951-01A1 (NIH)
Record Dates: First submitted 2016-02-02; First posted 2016-02-10 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: AIDS Dementia Complex
Keywords: HIV; Dementia; Neuroimaging
MeSH Terms: conditions — AIDS Dementia Complex; Dementia | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HIV+ with neurocognitive disorder (Experimental): All subjects will receive neurocognitive testing. Subjects will have a brain MRI prior to drug infusion. A one-time ferumoxytol IV infusion will be given at a dose of 4mg Fe/kg up to a maximum of 510mg of elemental iron delivered at a rate of 1ml/sec. A second brain MRI will be completed post-infusion
  Interventions: Drug: Ferumoxytol
- HIV+ without neurocognitive impairment (Active Comparator): All subjects will receive neurocognitive testing. Subjects will have a brain MRI prior to drug infusion. A one-time ferumoxytol IV infusion will be given at a dose of 4mg Fe/kg up to a maximum of 510mg of elemental iron delivered at a rate of 1ml/sec. A second brain MRI will be completed post-infusion
  Interventions: Drug: Ferumoxytol
- HIV- without neurocognitive impairment (Active Comparator): All subjects will receive neurocognitive testing. Subjects will have a brain MRI prior to drug infusion. A one-time ferumoxytol IV infusion will be given at a dose of 4mg Fe/kg up to a maximum of 510mg of elemental iron delivered at a rate of 1ml/sec. A second brain MRI will be completed post-infusion
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol — All subjects will receive neurocognitive testing. Subjects will have a brain MRI prior to drug infusion. A one-time ferumoxytol IV infusion will be given at a dose of 4mg Fe/kg up to a maximum of 510mg of elemental iron delivered at a rate of 1ml/sec. A second brain MRI will be completed post-infusion
  Other Names: Feraheme

SUMMARY:
This project will investigate the ability of a novel MRI contrast agent to identify and quantitate ongoing monocyte/macrophage (M/MΦ)-mediated inflammation in the brains of HIV-infected individuals.

DETAILED DESCRIPTION:
HIV-associated neurocognitive disorders (HAND) continue to be prevalent despite effective combination antiretroviral therapy (cART) and have a significant impact on morbidity and quality of life. Monocytes/macrophages (M/MΦ) are believed to play a critical role in the pathogenesis of HAND. Neuroimaging HIV research has not focused on assessing M/MΦ-mediated inflammation in the brain. Currently, no neuroimaging modality exists that can define the extent of active inflammation due to M/MΦ in HAND either as a clinical diagnostic tool or to assist in defining objective improvement in clinical trials addressing HAND. Ferumoxytol is an ultra-small iron oxide MRI contrast agent avidly taken up by circulating M/MΦ. The investigators hypothesize that ferumoxytol-based imaging can identify ongoing inflammation due to perivascular M/MΦ which is believed to represent a key pathologic correlate of HAND.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-65 years
* Plasma HIV RNA < 48 copies/ml (HIV+ subjects only)
* On stable cART >= 1 year (HIV+ subjects only)
* Global neuropsychological (NP) score <-0.5 in at least one cognitive domain known to be affected by HIV (neurocognitively impaired subjects only)
* Documentation of negative HIV infection by an FDA approved test (HIV- subjects only)

Exclusion Criteria:

* Active substance use
* History of myocardial infarct or stroke
* Diabetes
* Chronic hepatitis C virus (HCV) infection
* Uncontrolled major affective disorder, active psychosis, central nervous system disease that affects the brain structure, or other uncontrolled chronic medical condition that in the opinion of the investigator may impact NP testing or the study outcome
* Psychoactive or other medications which may impact NP testing
* Factors that preclude MRI
* Known hypersensitivity to ferumoxytol
* History of laboratory measurements consistent with an iron overload syndrome
* Medical conditions that require frequent blood transfusions
* Taking oral iron supplements
* Elevated iron levels
* Any condition, which in the opinion of the investigator, would compromise the subject's ability to participate
* Multiple drug allergies that may pose a greater risk of anaphylaxis associated with ferumoxytol
* Pregnant, unwillingness to practice birth control, or breastfeeding
* Unable to give informed consent

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of abnormal MRIs | Change from Baseline MRI at 4-6 weeks post-infusion MRI
  The proportion of abnormal MRIs will be compared for each group.

SECONDARY OUTCOMES:
Change in quantitative susceptibility mapping (QSM) | Change from Baseline MRI at 4-6 weeks post-infusion MRI
  Use of QSM to quantitate ferumoxytol accumulation in the brain

CONTACTS AND LOCATIONS:
Overall Officials: Beau Nakamoto, MD, PhD, Principal Investigator — University of Hawaii
Locations (1):
- Hawaii Center for AIDS, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No